CLINICAL TRIAL: NCT05047419
Title: Using Mobile Health Approaches to Improve Asthma Treatment
Brief Title: Asthma in Pregnancy
Status: Completed | Type: Observational
Sponsor: Linnea Polgreen (Other)
Responsible Party: Sponsor-Investigator, Linnea Polgreen, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 202104290
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Asthma; Pregnancy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant Participants with Asthma: Participants will be asked to use peak flow meter each day from enrollment to 6 weeks post due date and send peak flow and FEV1 values to the research team via text message. Also, every 3 months participants will be asked to send in a PDF of the values from the peak flow meter app for the previous 7 days via email as a validation of the text message values.
- Not Pregnant Participants with Asthma: Participants will be asked to use peak flow meter each day from enrollment to 9 months and send peak flow and FEV1 values to the research team via text message. Also, every 3 months participants will be asked to send in a PDF of the values from the peak flow meter app for the previous 7 days via email as a validation of the text message values.

SUMMARY:
The long-term goal is to improve the care of patients with asthma. The overarching objective of this pilot grant is to test the feasibility, acceptability and potential clinical utility of deploying a mobile-health intervention to improve asthma surveillance.

DETAILED DESCRIPTION:
Asthma is a major cause of morbidity. Asthma is frequently underdiagnosed, and proven therapies are underused. Even among patients treated for asthma, adherence to treatment is often is suboptimal.

Adherence to asthma therapy depends not only on regular use of therapies, but also correct technique for inhaler use. To improve treatments, home-based interventions have been proposed. Many such solutions involve collecting patient data to motivate patients and alert providers to ongoing problems. Examples of proposed solutions include using an app to keep symptom and medication logs, using Fitbits to document physical limitations, and nighttime breathing sensors. Other proposals include using peak expiratory flow meters, portable spirometers, and portable oscillometry. While promising, most of these efforts have, to date, not expanded widely beyond research settings.

Asthma during pregnancy is especially important to treat. Uncontrolled asthma is associated with preeclampsia, low birth weight, and fetal death. For some patients asthma is less severe during pregnancy, but for others, asthma worsens. In addition, pregnant patients with asthma often decrease use of medication or stop therapy altogether. Many pregnant patients stop therapy due to worry about negative effects on the baby. In general, asthma therapy is safe for pregnant patients and the babies, and hypoxia is dangerous for both.

Despite the importance of asthma treatment during pregnancy, some healthcare providers do not encourage pregnant patients with asthma to continue with asthma treatment. Many providers do not feel qualified to educate and treat patients during pregnancy, and pregnant patients may not be adequately informed that asthma therapy is safe. Also, pregnant patients may minimize their symptoms if worried about the safety of therapies. Accordingly, collecting objective information from patients in the home environment could improve the health of pregnant patients and the babies. Home monitoring may be especially important for patients living in rural areas with limited access to healthcare.

Home measurements of asthma symptoms can supplement clinic visits. However, this approach requires disciplined follow-up on the part of both patients and the healthcare team. Patients are required to use peak flow meters and regularly share results with providers. In addition, healthcare providers need to act on the shared data.

The purpose of this study is to determine if patients with asthma (pregnant and not pregnant) will take daily measurements with a peak flow meter and return them to the research team.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and write in English or Spanish;
* Current patient at participating clinic;
* Diagnosis of asthma;
* Owns a smartphone capable of supporting Bluetooth-enabled peak flow meter.

Exclusion Criteria:

* 3rd trimester of pregnancy;
* Current prisoner status;
* Unable to provide own written informed consent.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant and Not Pregnant participants with an Asthma diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Comparison of Number of Peak Flow Measurements Received | 9 months
  Comparison of number of peak flow measurements received between pregnant and not pregnant groups.

CONTACTS AND LOCATIONS:
Overall Officials: Linnea Polgreen, PHD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loftus PA, Wise SK. Epidemiology of asthma. Curr Opin Otolaryngol Head Neck Surg. 2016 Jun;24(3):245-9. doi: 10.1097/MOO.0000000000000262. PMID 26977741
- [Background] Cloutier MM. Asthma management programs for primary care providers: increasing adherence to asthma guidelines. Curr Opin Allergy Clin Immunol. 2016 Apr;16(2):142-7. doi: 10.1097/ACI.0000000000000242. PMID 26849166
- [Background] Morton RW, Elphick HE, Craven V, Shields MD, Kennedy L. Aerosol Therapy in Asthma-Why We Are Failing Our Patients and How We Can Do Better. Front Pediatr. 2020 Jun 11;8:305. doi: 10.3389/fped.2020.00305. eCollection 2020. PMID 32656165
- [Background] Moran C, Doyle F, Sulaiman I, Bennett K, Greene G, Molloy GJ, Reilly RB, Costello RW, Mellon L. The INCATM (Inhaler Compliance AssessmentTM): A comparison with established measures of adherence. Psychol Health. 2017 Oct;32(10):1266-1287. doi: 10.1080/08870446.2017.1290243. Epub 2017 Feb 28. PMID 28276739
- [Background] Greiwe J, Nyenhuis SM. Wearable Technology and How This Can Be Implemented into Clinical Practice. Curr Allergy Asthma Rep. 2020 Jun 6;20(8):36. doi: 10.1007/s11882-020-00927-3. PMID 32506184
- [Background] Kouri A, Gupta S, Yadollahi A, Ryan CM, Gershon AS, To T, Tarlo SM, Goldstein RS, Chapman KR, Chow CW. Addressing Reduced Laboratory-Based Pulmonary Function Testing During a Pandemic. Chest. 2020 Dec;158(6):2502-2510. doi: 10.1016/j.chest.2020.06.065. Epub 2020 Jul 8. PMID 32652095
- [Background] Bousquet J, Arnavielhe S, Bedbrook A, Bewick M, Laune D, Mathieu-Dupas E, Murray R, Onorato GL, Pepin JL, Picard R, Portejoie F, Costa E, Fonseca J, Lourenco O, Morais-Almeida M, Todo-Bom A, Cruz AA, da Silva J, Serpa FS, Illario M, Menditto E, Cecchi L, Monti R, Napoli L, Ventura MT, De Feo G, Larenas-Linnemann D, Fuentes Perez M, Huerta Villabolos YR, Rivero-Yeverino D, Rodriguez-Zagal E, Amat F, Annesi-Maesano I, Bosse I, Demoly P, Devillier P, Fontaine JF, Just J, Kuna TP, Samolinski B, Valiulis A, Emuzyte R, Kvedariene V, Ryan D, Sheikh A, Schmidt-Grendelmeier P, Klimek L, Pfaar O, Bergmann KC, Mosges R, Zuberbier T, Roller-Wirnsberger RE, Tomazic P, Fokkens WJ, Chavannes NH, Reitsma S, Anto JM, Cardona V, Dedeu T, Mullol J, Haahtela T, Salimaki J, Toppila-Salmi S, Valovirta E, Gemicioglu B, Yorgancioglu A, Papadopoulos N, Prokopakis EP, Bosnic-Anticevich S, O'Hehir R, Ivancevich JC, Neffen H, Zernotti E, Kull I, Melen E, Wickman M, Bachert C, Hellings P, Palkonen S, Bindslev-Jensen C, Eller E, Waserman S, Sova M, De Vries G, van Eerd M, Agache I, Casale T, Dykewickz M, Naclerio RN, Okamoto Y, Wallace DV; MASK study group. MASK 2017: ARIA digitally-enabled, integrated, person-centred care for rhinitis and asthma multimorbidity using real-world-evidence. Clin Transl Allergy. 2018 Oct 25;8:45. doi: 10.1186/s13601-018-0227-6. eCollection 2018. PMID 30386555
- [Background] Huffaker MF, Carchia M, Harris BU, Kethman WC, Murphy TE, Sakarovitch CCD, Qin F, Cornfield DN. Passive Nocturnal Physiologic Monitoring Enables Early Detection of Exacerbations in Children with Asthma. A Proof-of-Concept Study. Am J Respir Crit Care Med. 2018 Aug 1;198(3):320-328. doi: 10.1164/rccm.201712-2606OC. PMID 29688023
- [Background] McLaughlin K, Foureur M, Jensen ME, Murphy VE. Review and appraisal of guidelines for the management of asthma during pregnancy. Women Birth. 2018 Dec;31(6):e349-e357. doi: 10.1016/j.wombi.2018.01.008. Epub 2018 Feb 21. PMID 29475603
- [Background] Bonham CA, Patterson KC, Strek ME. Asthma Outcomes and Management During Pregnancy. Chest. 2018 Feb;153(2):515-527. doi: 10.1016/j.chest.2017.08.029. Epub 2017 Sep 1. PMID 28867295
- [Background] Robijn AL, Murphy VE, Gibson PG. Recent developments in asthma in pregnancy. Curr Opin Pulm Med. 2019 Jan;25(1):11-17. doi: 10.1097/MCP.0000000000000538. PMID 30407268
- [Background] Labor S, Dalbello Tir AM, Plavec D, Juric I, Roglic M, Pavkov Vukelic J, Labor M. What is safe enough - asthma in pregnancy - a review of current literature and recommendations. Asthma Res Pract. 2018 Dec 27;4:11. doi: 10.1186/s40733-018-0046-5. eCollection 2018. PMID 30607253